CLINICAL TRIAL: NCT00018798
Title: Longitudinal Evaluation of Chronic Combat-Related PTSD
Brief Title: Post-Traumatic Stress Disorder (PTSD) Symptom Study
Status: Completed | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: MHBS-001-99F
Record Dates: First submitted 2001-07-03; First posted 2001-07-05 (Estimated); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: PTSD
Keywords: Combat-Related PTSD, Vietnam Veterans
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Bi-weekly telephone calls: 34 participants received bi-weekly telephone calls in addition to the annual reviews
- Annual review only: 23 participants received annual reviews only

SUMMARY:
The primary goals for this investigation are to quantify: (1) fluctuations in PTSD symptom reports when assessed at bi-weekly intervals; (2) change in PTSD symptoms associated with stressful life events; and (3) change in PTSD symptoms associated with perceived social support.

DETAILED DESCRIPTION:
The primary goals for this investigation are to quantify: (1) fluctuations in PTSD symptom reports when assessed at bi-weekly intervals; (2) change in PTSD symptoms associated with stressful life events; and (3) change in PTSD symptoms associated with perceived social support.

Despite increased sophistication in measurement of PTSD, little is known about the long-term longitudinal course of this disorder or the fluctuation of symptoms over time. Because previous studies have focused on the development and persistence of symptoms immediately following a stressor, the course of the chronic disorder has been largely unexplored. Although there is evidence of both persistence and fluctuation of PTSD symptom presentation in Vietnam veterans, little is known about how much and in what ways symptoms change over time. This investigation will increase understanding of the nature and extent of symptom fluctuation as well as the longitudinal course of PTSD as first steps in determining which variables affect that course and how clinicians might intervene to alter it.

Aversive life events may constitute one factor that influences the course of chronic PTSD. Researchers and clinicians have frequently hypothesized that stressful life events account for much of the variability in course of chronic PTSD; individuals with PTSD may have a compromised ability to cope with stressors, and such events may worsen existing symptoms. Social support is another variable thought to affect the course of post-trauma symptomatology. Support from other persons has been shown to both promote psychological health in general and to protect against psychological deterioration in times of stress. This investigation will examine aversive life events and perceived social support to determine their relationships over time to symptoms of PTSD.

ELIGIBILITY:
Inclusion Criteria:

1. Vietnam vets who served in combat
2. Diagnosis of current or lifetime PTSD

Excluded if severe psychosis, current diagnosis of acute substance dependence, if no stable residence in past 6 months

Exclusion Criteria:

Actively psychosis, currently suicidal or homicidal, without telephone access, or had experienced substance or alcohol abuse or dependence within the previous six months.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Vietnam combat veterans
Sampling Method: Non-Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2000-04-01 (Actual); Primary Completion 2004-04-01 (Actual); Study Completion 2005-04-01 (Actual)

PRIMARY OUTCOMES:
PTSD Checklist - Military Version | For past two weeks
  The PTSD Checklist-Military Version is a self-report questionnaire comprising 17 items corresponding to the 17 DSM-IV symptoms for PTSD. Respondents are instructed to specify the extent to which they have been bothered by each symptom during the past month on a Likert-type scale ranging from 1 - not at all to 5 = extremely. Weathers et al. (1993) reported a full scale internal consistency reliability (coefficient alpha) for the PCL-M of .97 and test-retest reliability (2- to 3-day interval) of .96.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara L. Niles, PhD, Principal Investigator — VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA
Locations (1):
- VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Temporal Associations Among Chronic PTSD Symptoms in U.S. Combat Veterans — https://pmc.ncbi.nlm.nih.gov/articles/PMC6785199/
- See also: Posttraumatic stress disorder symptomatology in Vietnam veterans before and after September 11 — https://pubmed.ncbi.nlm.nih.gov/14555871/